CLINICAL TRIAL: NCT03370133
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo- and Active Comparator-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab Compared to Placebo and an Active Comparator in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: BE VIVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0009; 2016-003425-42 (EudraCT Number)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Chronic Plaque Psoriasis; Psoriatic Arthritis
Keywords: Bimekizumab; PSO; Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — bimekizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bimekizumab cohort (Experimental): Subjects will receive bimekizumab for 52 weeks.
  Interventions: Drug: Bimekizumab
- Ustekinumab cohort (Active Comparator): Subjects will receive ustekinumab (dose 1 or dose 2 depending on subjects weight) for 52 weeks. Placebo will be administered at pre-specified time points to maintain the blinding.
  Interventions: Drug: Ustekinumab; Other: Placebo
- Placebo (Placebo Comparator): Subjects will receive placebo up to week 16 and bimekizumab starting at week 16 through week 52.
  Interventions: Drug: Bimekizumab; Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab will be provided at pre-specified time intervals.
  Other Names: UCB4940
  Arms: Bimekizumab cohort; Placebo
Drug: Ustekinumab — Ustekinumab will be provided as dose 1 for subjects weighing <=100 kg and as dose 2 for subjects weighing >100 kg at pre-specified time intervals.
  Other Names: Stelara®
  Arms: Ustekinumab cohort
Other: Placebo — Subjects will receive Placebo at pre-specified time points.
  Other Names: PBO
  Arms: Placebo; Ustekinumab cohort

SUMMARY:
This is a study to compare the efficacy of bimekizumab versus placebo and an active comparator in the treatment of subjects with moderate to severe chronic plaque psoriasis (PSO).

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Chronic plaque psoriasis (PSO) for at least 6 months prior to the Screening Visit
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Investigator's Global Assessment (IGA) score >=3 on a 5-point scale
* Subject is a candidate for systemic PSO therapy and/or phototherapy
* Female subject of child bearing potential must be willing to use highly effective method of contraception

Exclusion Criteria:

* Subject has an active infection (except common cold), a recent serious infection, or a history of opportunistic or recurrent chronic infections
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any other condition, including medical or psychiatric, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study
* Presence of active suicidal ideation or positive suicide behavior
* Presence of moderately severe major depression or severe major depression
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (105):
- United States (25):
  - Ps0009 946, Phoenix, Arizona
  - Ps0009 910, Bakersfield, California
  - Ps0009 919, San Diego, California
  - Ps0009 906, Boca Raton, Florida
  - Ps0009 909, Boynton Beach, Florida
  - Ps0009 912, Coral Gables, Florida
  - Ps0009 907, Miami, Florida
  - Ps0009 903, Ocala, Florida
  - Ps0009 921, Ormond Beach, Florida
  - Ps0009 918, Tampa, Florida
  - Ps0009 941, Alpharetta, Georgia
  - Ps0009 911, Plainfield, Indiana
  - Ps0009 900, West Des Moines, Iowa
  - Ps0009 905, Overland Park, Kansas
  - Ps0009 922, Baton Rouge, Louisiana
  - Ps0009 917, Troy, Michigan
  - Ps0009 915, St Louis, Missouri
  - Ps0009 958, Omaha, Nebraska
  - Ps0009 901, Portsmouth, New Hampshire
  - Ps0009 908, East Windsor, New Jersey
  - Ps0009 923, Albuquerque, New Mexico
  - Ps0009 913, New York, New York
  - Ps0009 920, Portland, Oregon
  - Ps0009 924, Houston, Texas
  - Ps0009 914, San Antonio, Texas
- Australia (4):
  - Ps0009 004, Fremantle
  - Ps0009 005, Phillip
  - Ps0009 002, Westmead
  - Ps0009 009, Woolloongabba
- Belgium (3):
  - Ps0009 050, Brussels
  - Ps0009 052, Liège
  - Ps0009 051, Loverval
- Canada (6):
  - Ps0009 673, Halifax
  - Ps0009 652, Oakville
  - Ps0009 651, Richmond Hill
  - Ps0009 650, Surrey
  - Ps0009 653, Toronto
  - Ps0009 657, Waterloo
- Germany (10):
  - Ps0009 218, Bonn
  - Ps0009 209, Darmstadt
  - Ps0009 214, Erlangen
  - Ps0009 208, Frankfurt am Main
  - Ps0009 210, Friedrichshafen
  - Ps0009 211, Hamburg
  - Ps0009 212, Heidelberg
  - Ps0009 213, Mahlow
  - Ps0009 205, Osnabrück
  - Ps0009 217, Schweinfurt
- Hungary (4):
  - Ps0009 254, Budapest
  - Ps0009 255, Budapest
  - Ps0009 253, Orosháza
  - Ps0009 259, Szekszárd
- Italy (2):
  - Ps0009 300, Roma
  - Ps0009 303, Roma
- Japan (30):
  - Ps0009 629, Asahikawa
  - Ps0009 605, Bunkyō City
  - Ps0009 607, Chiyoda City
  - Ps0009 610, Chūōku
  - Ps0009 601, Fukuoka
  - Ps0009 619, Gifu
  - Ps0009 620, Hamamatsu
  - Ps0009 608, Itabashi-Ku
  - Ps0009 627, Itabashi-Ku
  - Ps0009 609, Kobe
  - Ps0009 600, Kurume
  - Ps0009 622, Matsumoto
  - Ps0009 604, Minatoku
  - Ps0009 623, Morioka
  - Ps0009 621, Nagoya
  - Ps0009 625, Nankoku
  - Ps0009 624, Obihiro
  - Ps0009 611, Osaka
  - Ps0009 614, Osaka
  - Ps0009 603, Sapporo
  - Ps0009 617, Sendai
  - Ps0009 613, Shimotsuke
  - Ps0009 602, Shinagawa-Ku
  - Ps0009 612, Shinjuku-Ku
  - Ps0009 618, Shinjuku-Ku
  - Ps0009 626, Shinjuku-Ku
  - Ps0009 628, Shinjuku-Ku
  - Ps0009 615, Sumida City
  - Ps0009 606, Takaoka
  - Ps0009 616, Tsu
- Poland (11):
  - Ps0009 362, Bialystok
  - Ps0009 369, Bialystok
  - Ps0009 371, Bydgoszcz
  - Ps0009 358, Katowice
  - Ps0009 357, Kielce
  - Ps0009 372, Lodz
  - Ps0009 374, Poznan
  - Ps0009 350, Warsaw
  - Ps0009 351, Warsaw
  - Ps0009 367, Wroclaw
  - Ps0009 370, Wroclaw
- Russia (4):
  - Ps0009 400, Moscow
  - Ps0009 402, Moscow
  - Ps0009 403, Moscow
  - Ps0009 404, Saint Petersburg
- United Kingdom (6):
  - Ps0009 556, Cardiff
  - Ps0009 551, Dundee
  - Ps0009 553, Edgbaston
  - Ps0009 552, Liverpool
  - Ps0009 550, Manchester
  - Ps0009 555, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asahina A, Okubo Y, Morita A, Tada Y, Igarashi A, Langley RG, Deherder D, Matano M, Vanvoorden V, Wang M, Ohtsuki M, Nakagawa H. Bimekizumab Efficacy and Safety in Japanese Patients with Plaque Psoriasis in BE VIVID: A Phase 3, Ustekinumab and Placebo-Controlled Study. Dermatol Ther (Heidelb). 2023 Mar;13(3):751-768. doi: 10.1007/s13555-022-00883-y. Epub 2023 Jan 17. PMID 36648594
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Rosmarin D, Lebwohl M, Peterson L, Madden C, de Cuyper D, Davies O, Thaci D. Bimekizumab safety in patients with moderate-to-severe plaque psoriasis: pooled data from up to 3 years of treatment in randomized phase III trials. Br J Dermatol. 2024 Mar 15;190(4):477-485. doi: 10.1093/bjd/ljad429. PMID 37950894
- [Result] Strober B, Boehncke WH, Krueger JG, Magnolo N, Vender R, Warren RB, Lopez Pinto JM, Kavanagh S, Hoepken B, Gisondi P. Bimekizumab Efficacy in Psoriasis by Subgroups: Post Hoc Analysis of Phase 3/3b Clinical Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3633-3650. doi: 10.1007/s13555-025-01557-1. Epub 2025 Oct 8. PMID 41060492
- [Result] Armstrong A, Papp KA, Lebwohl M, Savage LJ, Yamanaka K, Vlase DE, Warham R, Lambert J, Lopez Pinto JM, Wixted K, Thaci D. Bimekizumab Impact on Patient-Reported Outcomes in Plaque Psoriasis: 4-Year Results from BE SURE, BE VIVID, BE READY, and BE BRIGHT. Dermatol Ther (Heidelb). 2025 Dec 8. doi: 10.1007/s13555-025-01595-9. Online ahead of print. PMID 41359217
- [Derived] Merola JF, Warren RB, Thaci D, Gordon KB, Nishida E, Strober B, Conrad C, Kavanagh S, Lopez Pinto JM, Hoepken B, Gisondi P. Bimekizumab Complete Clearance of Both Skin and Nail Psoriasis: Comparative Efficacy in Phase III/IIIb Studies. Am J Clin Dermatol. 2025 Nov;26(6):967-979. doi: 10.1007/s40257-025-00968-2. Epub 2025 Aug 31. PMID 40886218
- [Derived] Merola JF, Gottlieb AB, Pinter A, Elewski B, Gooderham M, Warren RB, Piaserico S, Wixted K, Cross N, Tilt N, Wiegratz S, Mrowietz U. Bimekizumab Efficacy in High-Impact Areas: Pooled 2-Year Analysis in Scalp, Nail, and Palmoplantar Psoriasis from Phase 3/3b Randomized Controlled Trials. Dermatol Ther (Heidelb). 2024 Dec;14(12):3291-3306. doi: 10.1007/s13555-024-01295-w. Epub 2024 Nov 22. PMID 39578348
- [Derived] Kokolakis G, Warren RB, Strober B, Blauvelt A, Puig L, Morita A, Gooderham M, Korber A, Vanvoorden V, Wang M, de Cuyper D, Madden C, Nunez Gomez N, Lebwohl M. Bimekizumab efficacy and safety in patients with moderate-to-severe plaque psoriasis who switched from adalimumab, ustekinumab or secukinumab: results from phase III/IIIb trials. Br J Dermatol. 2023 Feb 22;188(3):330-340. doi: 10.1093/bjd/ljac089. PMID 36751950
- [Derived] Warren RB, Gottlieb AB, Merola JF, Garcia L, Cioffi C, Peterson L, Pelligra C, Ciaravino V. Psychometric Validation of the Psoriasis Symptoms and Impacts Measure (P-SIM), a Novel Patient-Reported Outcome Instrument for Patients with Plaque Psoriasis, Using Data from the BE VIVID and BE READY Phase 3 Trials. Dermatol Ther (Heidelb). 2021 Oct;11(5):1551-1569. doi: 10.1007/s13555-021-00570-4. Epub 2021 Jul 14. PMID 34260044
- [Derived] Reich K, Papp KA, Blauvelt A, Langley RG, Armstrong A, Warren RB, Gordon KB, Merola JF, Okubo Y, Madden C, Wang M, Cioffi C, Vanvoorden V, Lebwohl M. Bimekizumab versus ustekinumab for the treatment of moderate to severe plaque psoriasis (BE VIVID): efficacy and safety from a 52-week, multicentre, double-blind, active comparator and placebo controlled phase 3 trial. Lancet. 2021 Feb 6;397(10273):487-498. doi: 10.1016/S0140-6736(21)00125-2. PMID 33549193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll participants in December 2017 and concluded in December 2019.
Pre-assignment Details: The study included a 2-5 week Screening Period, a 16-week Initial Period and a 36-week Maintenance Period. After the Maintenance Period participants either enrolled in an open-label study or had a SFU Visit 20 weeks after their final dose (including those withdrawn from IMP). Participant Flow refers to the Randomized Set and Maintenance Set.
Groups:
- Placebo: Participants received placebo up to Week 16 and bimekizumab starting at Week 16 through Week 52.
- Bimekizumab (BKZ) 320 Milligrams (mg) Q4W: Participants received bimekizumab 320 mg Q4W for 52 weeks.
- Ustekinumab (Uste): Participants received ustekinumab 45 mg or 90 mg (depending on participants weight) for 52 weeks. Placebo was administered at pre-specified time points to maintain the blinding.
- Placebo/Bimekizumab 320 mg Q4W: After the 16-week Initial Treatment Period (Initial Period) participants initially randomized to placebo received bimekizumab 320 mg Q4W during the 36-week Maintenance Treatment Period (Maintenance Period).
- Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W: After the 16-week Initial Treatment Period participants initially randomized to bimekizumab 320 mg Q4W continued to receive bimekizumab 320 mg Q4W during the 36-week Maintenance Treatment Period.
- Ustekinumab/Ustekinumab: After the 16-week Initial Treatment Period participants initially randomized to ustekinumab 45 mg or 90 mg (depending on participant weight) continued to receive ustekinumab during the 36-week Maintenance Treatment Period.
Period: Initial Treatment Period (WK 16)
Arm/Group | Placebo | Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | Ustekinumab (Uste) | Placebo/Bimekizumab 320 mg Q4W | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W | Ustekinumab/Ustekinumab
Started | 83 | 321 | 163 | 0 | 0 | 0
Completed | 74 | 306 | 157 | 0 | 0 | 0
Not Completed | 9 | 15 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 5 | 2 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Site closed | 0 | 2 | 0 | 0 | 0 | 0
Period: Maintenance Treatment Period (WK 52)
Arm/Group | Placebo | Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | Ustekinumab (Uste) | Placebo/Bimekizumab 320 mg Q4W | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W | Ustekinumab/Ustekinumab
Started | 0 | 0 | 0 | 74 | 306 | 157
Completed | 0 | 0 | 0 | 69 | 283 | 141
Not Completed | 0 | 0 | 0 | 5 | 23 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 12 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4 | 4
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Consent Withdrawn for IMP Not Procedures | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Randomized Set (RS) consisting of all participants randomized into the study.
Arm/Group | Placebo | Bimekizumab (BKZ) 320 Milligrams (mg) Q4W | Ustekinumab (Uste) | Total Title
Number analyzed (Participants) | 83 | 321 | 163 | 567
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 1 | 3
  Between 18 and 65 years | 73 | 285 | 144 | 502
  >=65 years | 10 | 34 | 18 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (13.6) | 45.2 (14.0) | 46.0 (13.6) | 46.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 92 | 46 | 161
  Male | 60 | 229 | 117 | 406
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 0 | 1 | 1 | 2
  Asian | 20 | 71 | 36 | 127
  Black | 0 | 9 | 3 | 12
  White | 63 | 237 | 120 | 420
  Other/mixed | 0 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI90) Response at Week 16
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (RS): Participants received placebo up to Week 16 and bimekizumab 320 mg Q4W starting at Week 16 through Week 52. Participants formed the Randomized Set (RS).
- Bimekizumab 320 mg Q4W (RS): Participants received bimekizumab 320 mg Q4W for 52 weeks. Participants formed the RS.
- Ustekinumab (RS): Participants received ustekinumab 45 mg or 90 mg (depending on participants weight) for 52 weeks. Placebo was administered at pre-specified time points to maintain the blinding. Participants formed the RS.
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 4.8 | 85.0 | 49.7
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); Odds ratio was calculated using stratified CMH (Cochran-Mantel-Haenszel) test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups (BKZ 320 mg Q4W vs PBO) were based on the CMH test from the general association; Odds Ratio (OR) = 99.869, 95% CI 2-sided [34.020 to 293.175]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups (BKZ 320 mg Q4W vs Ustekinumab) were based on the CMH test from the general association; Odds Ratio (OR) = 6.056, 95% CI 2-sided [3.874 to 9.466]

2. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) (Clear or Almost Clear With at Least a 2-category Improvement From Baseline) Response at Week 16
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline at Week 16.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 4.8 | 84.1 | 53.4
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 118.762, 95% CI 2-sided [36.701 to 384.307]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.809, 95% CI 2-sided [3.096 to 7.470]

3. Secondary Outcome: Percentage of Participants With a PASI100 Response at Week 16
Description: The PASI100 response assessments are based on a 100% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 0 | 58.6 | 20.9
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); Odds ratio was calculated using stratified CMH test with region and prior biologic exposure as stratification variables. Logit method was used where CMH test not possible due to very low response; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 25.590, 95% CI 2-sided [9.063 to 72.253]

4. Secondary Outcome: Percentage of Participants With an IGA 0 Response at Week 16
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0] with at least a two-category improvement from Baseline at Week 16.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 0 | 58.6 | 22.1
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 25.471, 95% CI 2-sided [9.020 to 71.925]

5. Secondary Outcome: Percentage of Participants With a PASI75 Response at Week 4
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 4
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 2.4 | 76.9 | 15.3
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 123.020, 95% CI 2-sided [29.394 to 514.862]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); Odds ratio was calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 18.202, 95% CI 2-sided [10.998 to 30.123]

6. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary Response for Pain at Week 16
Description: As Patient-Reported-Outcome (PRO) measure, the PSD (further published as P-SIM) was used to assess key symptoms relevant to patients with moderate to severe plaque psoriasis. Site staff trained participants on the use of the electronic device used to collect ePRO diary data at Screening, device was then dispensed to the participant for home use until Week 16 Visit. The ePRO diary was completed on daily basis from Screening to Week 16 Visit.
  PSD pain item was assessed daily on a numeric rating scale (NRS) from 0 (no pain) to 10 (very severe pain). PSD score for pain at a given visit was an average of daily values over the week prior to the visit. The response was defined as an improvement (decrease) in pain score higher than the prespecified 1.98 response threshold at Week 16. The endpoint was characterized as percentage of participants with PSD pain response.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants. Number of participants analyzed reflect those with a Baseline score at or above the 1.98 response threshold.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 54 | 229 | 107
percentage of participants | 16.7 | 77.3 | 68.2
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 16.258, 95% CI 2-sided [7.356 to 35.931]

7. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary Response for Itch at Week 16
Description: A PRO measure, the PSD (further published as P-SIM) was used to assess key symptoms relevant to patients with moderate to severe plaque psoriasis. Site staff trained participants on the use of the electronic device used to collect ePRO diary data at Screening, device was then dispensed to participant for home use until Week 16 Visit. The ePRO diary was completed on daily basis from Screening to Week 16 Visit.
  PSD itch item was assessed daily on a NRS from 0 (no itch) to 10 (very severe itch). PSD score for itch was an average of daily values over the week prior to the visit. The response was defined as an improvement (decrease) in itch score higher than the prespecified 2.39 response threshold at Week 16. The endpoint was characterized as percentage of participants with a PSD itch response.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants. Number of participants analyzed reflect those with a Baseline score at or above the 2.39 response threshold.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 61 | 244 | 117
percentage of participants | 13.1 | 76.6 | 65.8
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 22.279, 95% CI 2-sided [9.795 to 50.674]

8. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary Response for Scaling at Week 16
Description: As PRO measure, the PSD (further published as P-SIM) was used to assess key symptoms relevant to patients with moderate to severe plaque psoriasis. Site staff trained participants on the use of the electronic device used to collect ePRO diary data at Screening, device was then dispensed to the participant for home use until Week 16 Visit. The ePRO diary was completed on daily basis from Screening to Week 16 Visit. PSD scaling item was assessed daily on a NRS from 0 (no scaling) to 10 (very severe scaling). PSD score for scaling was an average of daily values over the week prior to the visit. The response was defined as an improvement (decrease) in scaling score higher than the prespecified 2.86 response threshold at Week 16. The endpoint was characterized as percentage of participants with a PSD scaling response.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants. Number of participants analyzed reflect those with a Baseline score at or above the 2.86 response threshold.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 63 | 246 | 116
percentage of participants | 12.7 | 78.5 | 59.5
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 23.049, 95% CI 2-sided [10.201 to 52.077]

9. Secondary Outcome: Percentage of Participants With a Scalp IGA Response (Clear or Almost Clear) at Week 16 for Participants With Scalp Psoriasis (PSO) >=2 at Baseline
Description: Only participants with scalp involvement at Baseline completed the scalp IGA. Participants with scalp involvement at Baseline were defined as those with a scalp IGA score >0 at Baseline. Scalp lesions were assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale (0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4= Severe). Scalp IGA 0/1 response at Week 16 was defined as clear (0) or almost clear (1) with at least a 2-category improvement from Baseline to Week 16.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants. Number of participants analyzed reflect those with a Baseline score of at least 2.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 72 | 285 | 146
percentage of participants | 15.3 | 84.2 | 70.5
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 37.696, 95% CI 2-sided [16.920 to 83.987]

10. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 2.4 | 85.0 | 43.6
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); Odds ratio was calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 8.047, 95% CI 2-sided [5.107 to 12.679]

11. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: The Randomized Set (RS) consisted of all randomized study participants. Placebo was only provided up to Week 16 and was not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 321 | 163
percentage of participants | 81.9 | 55.8
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); Odds ratio was calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.795, 95% CI 2-sided [2.442 to 5.899]

12. Secondary Outcome: Percentage of Participants With an IGA (Clear or Almost Clear With at Least a 2-category Improvement From Baseline) Response at Week 12
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline at Week 12.
Time Frame: Week 12
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 83 | 321 | 163
percentage of participants | 4.8 | 81.9 | 52.1
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); Odds ratio was calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.379, 95% CI 2-sided [2.850 to 6.730]

13. Secondary Outcome: Percentage of Participants With an IGA (Clear or Almost Clear With at Least a 2-category Improvement From Baseline) Response at Week 52
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline at Week 52.
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W (RS) | Ustekinumab (RS)
Number analyzed (Participants) | 321 | 163
percentage of participants | 78.2 | 60.7
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Ustekinumab (RS); Odds ratio was calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.412, 95% CI 2-sided [1.573 to 3.699]

14. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) Adjusted by Duration of Subject Exposure to Study Treatment During the Initial Treatment Period
Description: The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the Adverse Event (AE) being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to end of Initial Treatment Period, including the Safety Follow-Up visit for those withdrawn from IMP (up to 36 weeks)
Population: The Safety Set (SS) consisted of all study participants that received at least 1 dose of IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Placebo (SS): Participants received placebo up to Week 16 and bimekizumab 320 mg Q4W starting at Week 16 through Week 52. Participants formed the Safety Set (SS).
- Bimekizumab 320 mg Q4W (SS): Participants received bimekizumab 320 mg Q4W for 52 weeks. Participants formed the SS.
- Ustekinumab (SS): Participants received ustekinumab 45 mg or 90 mg (depending on participants weight) for 52 weeks. Placebo was administered at pre-specified time points to maintain the blinding. Participants formed the SS.
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS) | Ustekinumab (SS)
Number analyzed (Participants) | 83 | 321 | 163
no. of new events per 100 subject-years | 238.41 [169.53 to 325.91] | 287.26 [246.93 to 332.29] | 247.62 [197.23 to 306.96]

15. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Subject Exposure to Study Treatment During the Initial Treatment Period
Description: The number of SAEs adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: as for outcome 14
Population: The Safety Set (SS) consisted of all study participants that received at least 1 dose of IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS) | Ustekinumab (SS)
Number analyzed (Participants) | 83 | 321 | 163
no. of new events per 100 subject-years | 7.97 [0.97 to 28.80] | 5.06 [1.64 to 11.80] | 10.14 [3.29 to 23.66]

16. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Subject Exposure to Study Treatment During the Initial Treatment Period
Description: The number of TEAEs leading to discontinuation adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: as for outcome 14
Population: The Safety Set (SS) consisted of all study participants that received at least 1 dose of IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS) | Ustekinumab (SS)
Number analyzed (Participants) | 83 | 321 | 163
no. of new events per 100 subject-years | 24.39 [8.95 to 53.09] | 6.08 [2.23 to 13.24] | 5.99 [1.24 to 17.52]

17. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) Adjusted by Duration of Subject Exposure to Study Treatment During the Maintenance Treatment Period
Description: The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the Adverse Event (AE) being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Week 16 to Safety Follow-Up (up to 52 weeks duration)
Population: The Maintenance Set (MS) consisted of all study participants who had received at least 1 dose of active IMP (bimekizumab or ustekinumab) in the Maintenance Treatment Period.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Placebo/Bimekizumab 320 mg Q4W (MS): After the 16-week Initial Treatment Period participants initially randomized to placebo received bimekizumab 320 mg Q4W during the 36-week Maintenance Treatment Period. Participants formed the Maintenance Set (MS).
- Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W (MS): After the 16-week Initial Treatment Period participants initially randomized to bimekizumab 320 mg Q4W continued to receive bimekizumab 320 mg Q4W during the 36-week Maintenance Treatment Period. Participants formed the MS.
- Ustekinumab/Ustekinumab (MS): After the 16-week Initial Treatment Period participants initially randomized to ustekinumab 45 mg or 90 mg (depending on participants weight) continued to receive ustekinumab 45 mg or 90 mg (depending on participants weight) during the 36-week Maintenance Treatment Period. Participants formed the MS.
Arm/Group | Placebo/Bimekizumab 320 mg Q4W (MS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W (MS) | Ustekinumab/Ustekinumab (MS)
Number analyzed (Participants) | 74 | 306 | 157
no. of new events per 100 subject-years | 149.35 [114.24 to 191.85] | 127.84 [111.58 to 145.81] | 111.24 [90.80 to 134.91]

18. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Subject Exposure to Study Treatment During the Maintenance Treatment Period
Description: as for outcome 15
Time Frame: From Week 16 to Safety Follow-Up (up to 52 weeks duration)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo/Bimekizumab 320 mg Q4W (MS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W (MS) | Ustekinumab/Ustekinumab (MS)
Number analyzed (Participants) | 74 | 306 | 157
no. of new events per 100 subject-years | 9.88 [3.21 to 23.05] | 6.19 [3.30 to 10.58] | 7.46 [3.22 to 14.70]

19. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Subject Exposure to Study Treatment During the Maintenance Treatment Period
Description: as for outcome 16
Time Frame: From Week 16 to Safety Follow-Up (up to 52 weeks duration)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo/Bimekizumab 320 mg Q4W (MS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W (MS) | Ustekinumab/Ustekinumab (MS)
Number analyzed (Participants) | 74 | 306 | 157
no. of new events per 100 subject-years | 5.91 [1.22 to 17.27] | 5.72 [2.95 to 9.99] | 3.71 [1.01 to 9.51]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected from Baseline to Safety Follow Up (up to Week 68)
Description: Treatment-emergent AEs were defined as those AEs that had a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week Safety Follow-Up [SFU] Period). Deaths in Any bimekizumab 320 mg Q4W arm occurred in the Initial Period (1 in placebo/ 1 in bimekizumab 320 mg Q4W).
Groups:
- Placebo Initial Period (SS): During the 16-week Initial Treatment Period participants received placebo. Participants formed the Safety Set (SS).
- Bimekizumab 320 mg Q4W Initial Period (SS): During the 16-week Initial Treatment Period participants received bimekizumab 320 mg Q4W. Participants formed the SS.
- Ustekinumab Initial Period (SS): During the 16-week Initial Treatment Period participants received ustekinumab 45 mg or 90 mg (depending on participants weight). Participants formed the SS.
- Any Bimekizumab 320 mg Q4W (AMS): This arm consisted of all participants who received bimekizumab 320 mg Q4W at any time in the study (up to Week 52). It also includes the participants that switched from placebo to bimekizumab 320 mg Q4W after the 16-week Initial Treatment Period. Participants formed the SS.
- Any Ustekinumab (AMS): This arm consisted of all participants who received ustekinumab 45 mg or 90 mg (depending on participants weight) at any time in the study (up to Week 52). Participants formed the SS.
Arm/Group | Placebo Initial Period (SS) | Bimekizumab 320 mg Q4W Initial Period (SS) | Ustekinumab Initial Period (SS) | Any Bimekizumab 320 mg Q4W (AMS) | Any Ustekinumab (AMS)
All-Cause Mortality (participants affected / at risk) | 1/83 | 1/321 | 1/163 | 2/395 | 1/163
Serious Adverse Events (participants affected / at risk) | 2/83 | 5/321 | 5/163 | 24/395 | 13/163
Other Adverse Events (participants affected / at risk) | 17/83 | 87/321 | 37/163 | 192/395 | 73/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Initial Period (SS) (N=83) | Bimekizumab 320 mg Q4W Initial Period (SS) (N=321) | Ustekinumab Initial Period (SS) (N=163) | Any Bimekizumab 320 mg Q4W (AMS) (N=395) | Any Ustekinumab (AMS) (N=163)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subglottic laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
False positive tuberculosis test (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Initial Period (SS) (N=83) | Bimekizumab 320 mg Q4W Initial Period (SS) (N=321) | Ustekinumab Initial Period (SS) (N=163) | Any Bimekizumab 320 mg Q4W (AMS) (N=395) | Any Ustekinumab (AMS) (N=163)
Nasopharyngitis (Infections and infestations) | 7 (8) | 30 (35) | 14 (15) | 86 (121) | 36 (53)
Oral candidiasis (Infections and infestations) | 0 (0) | 28 (30) | 0 (0) | 60 (98) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 9 (9) | 5 (6) | 36 (48) | 18 (22)
Urinary tract infection (Infections and infestations) | 5 (5) | 6 (6) | 1 (1) | 12 (14) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 10 (10) | 9 (10)
Headache (Nervous system disorders) | 0 (0) | 11 (11) | 7 (10) | 16 (17) | 10 (14)
Psoriasis (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4) | 2 (2) | 9 (11) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 7 (7) | 5 (5) | 14 (14) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03370133/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03370133/SAP_001.pdf